CLINICAL TRIAL: NCT07321977
Title: Assessment of a Portable Digital Device for Quantified Analysis of Markerless Walking in Volunteers With Neuromuscular Diseases or Asymptomatic Volunteers
Acronym: Myokinesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Myokinesis
Record Dates: First submitted 2025-12-15; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy (SMA); Charcot-Marie-Tooth; Muscular Dystrophy; Myotonic Dystrophy
Keywords: gait analysis; neuromuscular; disease; markerless
MeSH Terms: conditions — Muscular Atrophy, Spinal; Charcot-Marie-Tooth Disease; Muscular Dystrophies; Myotonic Dystrophy; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers with Neuromuscular disease or asymptomatic (Other): All participants have the same intervention. The intervention is to walk with shoes in a gait analysis room with VICON markers on the body. At the same time, the participant will be film by two smartphones to compare the kinematics and the spatio-temporal parameters between a marker-based and a markerless gait analysis.
  Interventions: Other: Gait analysis via video capture

INTERVENTIONS:
Other: Gait analysis via video capture — Using motion analysis software integrated into a smartphone

SUMMARY:
In recent years, knowledge of neuromuscular diseases has advanced considerably, and new therapeutic avenues are beginning to emerge. The proliferation of clinical trials has created a need to identify biomarkers that are both sensitive to changes and specific to the disease. Current gait tests only consider the time factor and not the evolution of the patient's biomechanics, which may prove insufficient for patients whose symptoms generally progress slowly. Quantifying gait parameters in neuromuscular patients therefore appears necessary. This is why we propose to study markerless gait analysis in this population, which would allow for simple and effective monitoring of kinematic parameters without resorting to complex equipment incompatible with routine clinical practice.

ELIGIBILITY:
* All volunteers

  * Age between 18 and 65
  * Ambulatory
  * Informed consent to participate in the study
  * Member of or beneficiary of a social security system
* Volunteers with a neuromuscular disease

  * Confirmed diagnosis of a neuromuscular disease of genetic origin (medical document to be provided upon enrollment in the study with proof of diagnosis) belonging to the list above.
  * Ability to walk for 2 minutes without assistance.
  * Ability to stand up from a chair with armrests at least 3 times in 30 seconds.
  * Ability to climb an inclined plane independently or with assistance to access the movement analysis room.

Exclusion Criteria

* All volunteers

  * Individuals under guardianship, curatorship, or legal protection
  * Pregnant or breastfeeding women
  * Non-ambulatory individuals
  * Individuals with epilepsy
  * Skin conditions preventing the placement of VICON motion sensors
* Asymptomatic volunteers

  * Unstable respiratory or cardiac problems
  * Neurological, musculoskeletal, or psychiatric problems
* Volunteers with a neuromuscular disease

  * Recent trauma or serious falls (≤ 6 months)
  * Individuals who have fallen more than twice in the past year and at least once in the past three months
  * Use of assistive devices such as rigid knee braces or walkers
  * Unstable cardiomyopathy
  * Individuals awaiting diagnosis

Exclusion criteria

* Inability to comply with the protocol requirements
* Medical or social conditions that could interfere with the study, as determined by the coordinating investigator or co-investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-07-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Vicon vs Myokinesis system correlation coefficient | Day 1
  Correlation coefficient between measurements from the two systems in both groups, for spatiotemporal parameters and joint range of motion in the sagittal plane at the hip, knee, and ankle

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Exploration et d'Évaluation Neuromusculaire, Paris, France